CLINICAL TRIAL: NCT06440681
Title: Effects of a 6-month Lifestyle Intervention Program in the DNAm PhenoAge, SOST, and GDF15 Markers of Biological Aging in Adults With Prediabetes
Brief Title: Effects of Lifestyle Intervention in the Biological Aging in Prediabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Ahmed Shafi Alenezi, Principle Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB log Number:2024-8
Record Dates: First submitted 2024-05-20; First posted 2024-06-04 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: PreDiabetes; Marker; Structural
Keywords: DNAm PhenoAge; Lifestyle modification; SOST; DGF-15
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: A 6-month lifestyle modification program will be launched at primary health centers in Arar, Saudi Arabia. 500 participants will be involved and all participants will be advised to: Reducing weight (5% of the basic weight), Exercise (4 hours/week), Moderate fat consumption (total fat 30% of total energy intake and saturated fat 10%). % of total energy consumed), A diet rich in fiber (15 g/1000 calories). Participants will receive individual, detailed, ongoing nutritional counseling by the study dietitian every two weeks. They will also be encouraged to participate in physical activities. The table below shows the detailed intervention for both groups.
  Finally, the participants will be divided into two groups:
  Lifestyle Modification Group (LMP): those who agreed and followed the previous instructions and advice. Control group (CG): those who did not receive health education or did not follow previous instructions or advice.
Who Masked: Participant
Masking Description: There is nothing masked to study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Modification Group (LMP) (Active Comparator): They are the people who will follow the lifestyle modification program, which is:
  Dietary counseling and monitoring: reduce fat intake (30% of total energy and saturated fat 10% of total energy) and increase fiber intake (15 g/1000 kcal) in the diet Physical activity: moderate exercise (150 minutes/week)
  Interventions: Other: Providing nutritional counselling; Other: counseling on physical activity
- Control group (CG) (Placebo Comparator): They are people who will not follow the lifestyle modification program or they did not know about this program
  Interventions: Other: Providing nutritional counselling; Other: counseling on physical activity

INTERVENTIONS:
Other: Providing nutritional counselling — Dietary counseling and monitoring:
  Reduce fat intake (30% of total energy and saturated fat 10% of total energy) and increase fiber intake (15 g/1000 kcal) in the diet.
  Participants will receive individual, detailed, ongoing nutritional counseling by the study dietitian every two weeks.
Other: counseling on physical activity — Physical activity:
  Participants will also be encouraged to participate in physical activities. moderate exercise (150 minutes/week)

SUMMARY:
Lifestyle modifications, including dietary changes and increased physical activity, play a crucial role in controlling complications to reduce or eliminate them. As well as controlling disturbances in biochemical markers such as DNAm PhenoAge, and signs of aging such as circulating sclerostin (SOST) and growth differentiation factor 15 (GDF15). This study seeks to address this dilemma by focusing on specific groups of elderly Saudis with prediabetes . Lifestyle changes in elderly Saudis with prediabetes show promise in reducing or eliminating complications. The potential insights derived from this research extend beyond academia, offering tangible benefits for clinical practice and public health

The proposed study will be implemented to achieve the following objective:

1. To determine changes in DNAm PhenoAge of elderly Saudis with prediabetes who underwent a 6-month lifestyle modification program.
2. To determine changes in other candidate senescence markers such as circulating sclerostin (SOST) and growth differentiation factor 15 (GDF15) of elderly Saudis with prediabetes who underwent a 6-month lifestyle modification program.

DETAILED DESCRIPTION:
Participants will be received at all healthcare centers in Arar, Kingdom of Saudi Arabia. They will be informed about the lifestyle modification intervention programme. The interview will take place in a designated and prepared place.

If approved, informed consent is signed. The procedures begin with filling out questionnaires and basic assessments include anthropometric, blood pressure and blood pressure measurements. The anthropometric measurements will be performed by well-trained medical staff. Height (m) and weight (kg) will be measured in light clothing without shoes. Waist, hip, circumference (cm) will be measured using a standard tape measure. BMI will be calculated by dividing weight in kilograms by the square of height in metres. Your blood pressure will be measured at each visit after adequate rest.

Dietary intake will be assessed through a validated food frequency questionnaire. Assessments will be repeated twice (at baseline and 6 months) in both groups. Fasting blood samples will then be collected using a sterile blood collection device to perform blood tests for biological age using self-analyzers in the internal laboratory of the participating primary health care centers. Tests will include complete blood count, serum albumin, creatinine, fasting glucose, C-reactive protein, alkaline phosphatase and other markers of aging such as SOST and DGF-15. Through these tests, the DNAm PhenoAge will be calculated through an online platform (https://thrivous.com/pages/biological-age Calculator).

In light of the results, participants will be included or excluded, and participants included in the program will continue with us through follow-up with nutritional awareness. 500 participants will be involved and all participants will be advised to:

Weight loss (5% of basic weight), exercise (4 hours/week), moderate fat consumption, and a diet rich in fiber.

5- Participants will receive individual, detailed and ongoing nutritional counseling through the study dietitian every two weeks, and they will also be encouraged to participate in physical activities. Table The detailed intervention for both groups is shown below. The measurements and analyzes will be repeated a few months after the beginning, and based on this, the Lifestyle Modification Group (LMP) will be determined: those who agreed and followed the previous instructions and advice.

The control group (CG): They are those who did not receive health education or did not follow previous instructions or advice.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of pre-diabetes for all Saudis aged 30 years and above, males and females
2. They must be able to exercise and be able to follow a diet

Exclusion Criteria

1. Insulin-dependent diabetes and non-diabetic patients
2. People with diseases that prevent them from participating and doing exercises

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in the rate of measurements of Age marker Albumin post intervention | 6 months
  Change in Albumin (g/L)
Change in the rate of measurements of Age marker fasting glucose post intervention | 6 months
  Change in fasting glucose (mmol/L)
Change in the rate of measurements of Age marker Creatinine post intervention | 6 months
  Change in Creatinine (umol/L)
Change in the rate of measurements of Age marker C-Reactive Protein post intervention | 6 months
  Change in C-Reactive Protein (mg/dL)
Change in the rate of measurements of Age marker Alkaline Phosphatase post intervention | 6 months
  Change in Alkaline Phosphatase (U/L)
Change in the rate of measurements of Age marker White Blood Cell Count (WBC) post intervention | 6 months
  Change in White Blood Cell Count (WBC) (10^3/uL)
Change in the rate of measurements of Age marker Lymphocyte post intervention | 6 months
  Change in Lymphocyte (%)
Change in the rate of measurements of Age marker Mean Cell Volume (MCV) post intervention | 6 months
  Change in Mean Cell Volume (MCV) (fL)
Change in the rate of measurements of Age marker Red Cell Distribution Width (RDW) post intervention | 6 months
  Change in Red Cell Distribution Width (RDW) (%)

SECONDARY OUTCOMES:
Change in the rate of measurements of Age marker SOST post intervention | 6 months
  Change in SOST(pmol/L)
Change in the rate of measurements of Age marker GDF15 post intervention | 6 months
  Change in GDF15 (10^3 pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Shaun B Sabico, M.D.PhD, Study Chair — King Saud University

IPD SHARING:
Plan to Share IPD: No